CLINICAL TRIAL: NCT00939146
Title: Outlook: An Intervention to Improve Quality of Life in Serious Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00011193; 1P01NR010948-01 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure; Renal Disease
Keywords: self management; quality of life; end of life
MeSH Terms: conditions — Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure; Kidney Diseases; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outlook Attention Control (Other): Subjects in the relaxation meditation group will meet with a facilitator three times, for a period of forty-five minutes each; they will listen to a non-guided relaxation CD.
  Interventions: Other: Outlook Attention Control
- Outlook Intervention (Other): The Outlook intervention is designed to assist patients self-manage role changes by guiding them through life review, current issues of forgiveness and conflict resolution, and future orientation, with planning heritage and legacy.
  Interventions: Other: Outlook Intervention

INTERVENTIONS:
Other: Outlook Attention Control — Subjects in the relaxation meditation group will meet with a facilitator three times, for a period of forty-five minutes each; they will listen to a non-guided relaxation CD.
  Arms: Outlook Attention Control
Other: Outlook Intervention — The Outlook intervention is designed to assist patients self-manage role changes by guiding them through life review, current issues of forgiveness and conflict resolution, and future orientation, with planning heritage and legacy.
  Arms: Outlook Intervention

SUMMARY:
This study will demonstrate whether an end-of-life preparation and completion intervention reduces anxiety, depression, pain and other symptoms and improves functional status, spiritual well-being, and quality of life. If effective, the intervention offers a brief, inexpensive, and transportable non-physician treatment method for improving the experience of individuals in the latter stages of life-limiting illness.

DETAILED DESCRIPTION:
Efforts to improve end-of-care often focus on pain and symptom control, but few, if any, effective interventions exist addressing preparation and completion. We designed an end-of-life preparation and completion intervention, based on the human development literature identifying life completion as a developmental task and the robust evidence in health communication and clinical psychology that addresses the value of expressing emotions and stress on health outcomes. Our specific aims are 1) evaluate the impact of an intervention that promotes discussions of end-of-life preparation and completion on health outcomes in dying persons, including pain and symptoms, physical function, emotional function (anxiety and depression), spiritual well-being, and quality of life at the end of life and 2) evaluate the content of the such discussions, examining task variation associated with gender, ethnicity, socio-economic status, quality of communication with family, spirituality, and stage of illness to improve understanding of the need for tailored intervention content based on demographics or location in the trajectory of illness. We propose a randomized control trial to evaluate the intervention. 140 patients with advanced cancer, CHF, ESRD, or COPD will be randomly assigned into one of two intervention groups and complete a brief battery of pre-test measures. Subjects in the first group ("treatment") will meet with a facilitator three times for a period of forty-five minutes each. In the first session, subjects will be asked to discuss issues related to life review. A week later, participants will be asked to speak in more depth about issues such as regret, forgiveness and things left undone. In the final session, a week hence, subjects will focus on heritage and legacy. The subjects in the second group ("attention control") will meet with a facilitator three times for a period of forty-five minutes each and be asked to listen to a non-guided relaxation CD. One week and two weeks later, participants in all groups will receive post-test measures administered by a blinded interviewer.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must have advanced life-limiting illness as determined by clinical criteria indicative of advance disease. Must be diagnosed with one of the following:

* Cancer: Stage IV metastatic cancer, pancreatic and lung cancers may include Stages III and IV, recurrent/refractory disease (multiple myeloma and related cancers);
* Congestive Heart Failure: NYHA Class III or IV;
* End-Stage Renal Disease: Dialysis dependent;
* Chronic Obstructive Pulmonary Disease: Oxygen dependent.

Also, eligible patients must receive care for one of the diseases above at Duke University Medical Center, have access to a telephone, live within a 35-mile radius of Durham, be at least 18 years of age, English speaking, and cognitively capable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
QUAL-E subscale describing preparation for death (Quality of Life at End of Life, Steinhauser et al. 2004) | Eight weeks

SECONDARY OUTCOMES:
Remaining subscales of the QUAL-E instrument (Quality of Life at End of Life, Steinhauser et al. 2004) | Eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen Steinhauser, PhD, Principal Investigator — Duke University; James A Tulsky, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States